CLINICAL TRIAL: NCT03352973
Title: Regulation of Craving in Internet Gamers: Neural Mechanisms and tDCS Intervention
Brief Title: Regulation of Craving in Internet Gamers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, jintao, zhang, Associated Professor, Beijing Normal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IGDROC
Record Dates: First submitted 2017-11-13; First posted 2017-11-24 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: within-subject, sham-controlled design: all subjects will receive active and sham tDCS in a randomized order
Who Masked: Participant, Investigator
Masking Description: double blind: both participants and experiment won't know the stimulation condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS on the dlPFC (Experimental): tDCS on the DLPFC Dorsolateral prefrontal cortex (DLPFC) target will be identified by the baseline functional magnetic resonance imaging (fMRI) study for regulation of craving using a separate sample. During the intervention, each participant will receive an active transcranial direct current stimulation (tDCS) intervention on this DLPFC region (1.5 mA for 20 minutes).
  Interventions: Other: active tDCS on the dlPFC
- sham tDCS on the dlPFC (Sham Comparator): Each participant will also receive a sham tDCS intervention as a controlled condition. The sham tDCS only include a 30-s ramp up and a 30-s ramp down.
  Interventions: Other: sham tDCS on the dlPFC

INTERVENTIONS:
Other: active tDCS on the dlPFC — During active tDCS session, participants will perform the regulation of craving (ROC) and emotion regulation (ER) tasks. In the ROC task, participants will downregulate and upregulate craving elicited by gaming pictures using cognitive reappraisal. In the ER task, participants will downregulate and upregulate aversive feelings by negative pictures using cognitive reappraisal. After the active tDCS session, participants will complete a cognitive task assessing inhibitory control of attentional bias, in which participants will perform a number classification task with gaming pictures and non-gaming pictures being distractors. During the task, reaction times (RTs) wil be recorded.
  Other Names: tDCS
  Arms: active tDCS on the dlPFC
Other: sham tDCS on the dlPFC — During the sham tDCS session, participants will perform the regulation of craving (ROC) and emotion regulation (ER) tasks. In the ROC task, participants will downregulate and upregulate craving elicited by gaming pictures using cognitive reappraisal. In the ER task, participants will downregulate and upregulate aversive feelings by negative pictures using cognitive reappraisal. After the sham tDCS session, participants will complete a cognitive task assessing inhibitory control of attentional bias, in which participants will perform a number classification task with gaming pictures and non-gaming pictures being distractors. During the task, reaction times (RTs) wil be recorded.
  Other Names: tDCS
  Arms: sham tDCS on the dlPFC

SUMMARY:
This project aims to investigate (1) the behavioral and neural mechanisms of regulation of craving in Internet gamers; (2) effects of tDCS over the dorsal lateral prefrontal cortex (dlPFC) on craving and regulation of craving and aversive emotions in this population. (3) effects of tDCS over dlPFC on attentional bias towards gaming related cues.This project will be conducted in Beijing, China, based on a large sample of Internet gamers.

DETAILED DESCRIPTION:
As with the experiment about tDCS effects on regulation of craving and aversive emotions, the experiment aims to test whether tDCS over dlPFC will enhance cognitive regulation of craving and aversive emotions. It is a within-subject, sham-controlled, double-blind design. Each participant receive both active and sham tDCS of dlPFC in a randomized order separated by one week. During both active and sham tDCS sessions, participants will perform regulation of craving (ROC) and emotion regulation (ER) tasks. In the ROC task, participants will be asked to downregulate and upregulate craving elicited by gaming pictures using cognitive reappraisal. In the ER task, participants will be asked to downregulate and upregulate aversive feelings elicited by negative pictures using cognitive reappraisal. During these tasks, self-report ratings and skin conductance responses (SCRs) will be recorded. The cognitive regulation ability is indexed by rating and SCRs differences between the up- and downregulation conditions.

As with the experiment about tDCS effects on attentional bias, the experiment aims to test whether tDCS over dlPFC will enhance inhibitory control of attentional bias towards gaming related cues. The inhibitory control of attentional bias will be measured by a cognitive task in which participants will perform a number classification task with gaming pictures and non-gaming pictures being distractors. The experiment is a within-subject, sham-controlled, double-blind design. Each participant will receive both active and sham tDCS of dlPFC in a randomized order separated by one week. After each tDCS session, participants will complete the cognitive task assessing inhibitory control of attentional bias. During the task, reaction times (RTs) wil be recorded. The attentional bias is indexed by RTs differences between trials with gaming pictures and trials with non-gaming pictures.

ELIGIBILITY:
Inclusion Criteria:

* engagement in a popular Internet game (Arena of Valor) for over 14 hours per week for a minimum of 6 months.

Exclusion Criteria:

* current or history of use of illegal substances and gambling;
* current or history of psychiatric or neurological illness;
* current use of psychotropic medications.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-10-20 (Actual)

PRIMARY OUTCOMES:
Craving in the regulation of craving (ROC) task after the initiation of active and sham tDCS | 4 minutes after the initiation of active and sham tDCS for half of the participants
  Using the Visual Analog Scale (from 1 = 'not at all' to 9 = 'very much'), craving is assessed in the ROC task. This task lasts 12-13 minutes. Craving in the downregulation condition will be compared between the active and sham tDCS. Craving in the upregulation condition will also be compared between the active and sham tDCS.
Aversive feeling in the emotion regulation (ER) task after the initiation of active and sham tDCS | 16-17 minutes after the initiation of active and sham tDCS
  Using the Visual Analog Scale (from 1 = 'not at all' to 9 = 'very much'), aversive feeling is assessed in the ER task. This task lasts 12-13 minutes. Aversive feeling in the downregulation condition will be compared between the active and sham tDCS. Aversive feeling in the upregulation condition will also be compared between the active and sham tDCS.
Reaction times (RTs) in the cognitive task assessing inhibition of attentional bias after the initiation of active and sham tDCS | 45-47 minutes after the initiation of of active and sham tDCS
  Using the E-prime software, RTs are recorded in milliseconds in the cognitive task assessing inhibition of attentional bias. The cognitive task lasts 5-6 minutes. RTs difference between the trials including gaming pictures and those including gaming pictures will be calculated and such RTs difference will be compared between the active and sham tDCS.

SECONDARY OUTCOMES:
Skin conductance responses (SCRs) in the ROC task after the initiation of active and sham tDCS | 4 minutes after the initiation of active and sham tDCS
  Using a biosignal recorder, SCRs are recorded in μs in the ROC task. This task lasts 12-13 minutes. SCRs in the downregulation condition will be compared between the active and sham tDCS. SCRs in the upregulation condition will also be compared between the active and sham tDCS.
Skin conductance responses (SCRs) in the ER task after the initiation of active and sham tDCS | 16-17 minutes after the initiation of active and sham tDCS ham tDCS
  Using a biosignal recorder, SCRs are recorded in μs in the ER task. This task lasts 12-13 minutes. SCRs in the downregulation condition will be compared between the active and sham tDCS. SCRs in the upregulation condition will also be compared between the active and sham tDCS.
Background craving before the initiation of active and sham tDCS | Approximately 10 minutes before the initiation of active and sham tDCS
  Using the Visual Analog Scale (from 1 = 'not at all' to 9 = 'very much'), background craving is assessed with a one-item questionaire (how much do you crave playing internet games now?). This assessment lasts approximately 1 minute. Background craving will be compared between the active and sham tDCS.
Cue-induced craving before the initiation of active and sham tDCS | Approximately 8 minutes before the initiation of active and sham tDCS
  Using the Visual Analog Scale (from 1 = 'not at all' to 9 = 'very much'), cue-induced craving is assessed in a cue-reactivity task. This assessment lasts 1-2 minutes. Cue-induced craving will be compared between the active and sham tDCS.
Background craving after the initiation of active and sham tDCS | 38-40 minutes after the the initiation of active and sham tDCS
  Using the Visual Analog Scale (from 1 = 'not at all' to 9 = 'very much'), background craving is assessed with a one-item questionaire (how much do you crave playing internet games now?). This assessment lasts approximately 1 minute. Background craving will be compared between the active and sham tDCS.
Cue-induced craving after the initiation of active and sham tDCS | 40-42 minutes after the the initiation of active and sham tDCS
  Using the Visual Analog Scale (from 1 = 'not at all' to 9 = 'very much'), cue-induced craving is assessed in a cue-reactivity task. This assessment lasts 1-2 minutes. Cue-induced craving will be compared between the active and sham tDCS.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tao Zhang, PhD, Principal Investigator — Beijing Normal University
Locations (1):
- State Key Laboratory of Cognitive Neuroscience and Learning, Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kober H, Mende-Siedlecki P, Kross EF, Weber J, Mischel W, Hart CL, Ochsner KN. Prefrontal-striatal pathway underlies cognitive regulation of craving. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14811-6. doi: 10.1073/pnas.1007779107. Epub 2010 Aug 2. PMID 20679212
- [Derived] Wu LL, Potenza MN, Zhou N, Kober H, Shi XH, Yip SW, Xu JH, Zhu L, Wang R, Liu GQ, Zhang JT. Efficacy of single-session transcranial direct current stimulation on addiction-related inhibitory control and craving: a randomized trial in males with Internet gaming disorder. J Psychiatry Neurosci. 2021 Jan 4;46(1):E111-E118. doi: 10.1503/jpn.190137. PMID 33119491